CLINICAL TRIAL: NCT02076906
Title: Safety and Feasibility Study of Using MR-guided High Intensity Focused Ultrasound (HIFU) for the Ablation of Relapsed or Refractory Pediatric Solid Tumors
Brief Title: MR-guided High Intensity Focused Ultrasound (HIFU) on Pediatric Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AeRang Kim (Other)
Responsible Party: Sponsor-Investigator, AeRang Kim, MD, PhD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU Pediatric Solid Tumors
Record Dates: First submitted 2014-01-28; First posted 2014-03-04 (Estimated); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Relapsed Pediatric Solid Tumors; Refractory Pediatric Solid Tumors; Rhabdomyosarcoma; Ewing Sarcoma; Osteosarcoma; Neuroblastoma; Wilms Tumor; Hepatic Tumor; Germ Cell Tumor; Desmoid Tumor
Keywords: relapsed pediatric solid tumors; refractory pediatric solid tumors; high intensity focused ultrasound; rhabdomyosarcoma; Ewing's sarcoma; osteosarcoma; neuroblastoma; Wilms' tumor; hepatic tumors; germ cell tumors; desmoid tumor
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Ewing; Osteosarcoma; Neuroblastoma; Wilms Tumor; Carcinoma, Hepatocellular; Neoplasms, Germ Cell and Embryonal; Desmoid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-HIFU (Experimental): Magnetic Resonance High Intensity Focused Ultrasound (MR-HIFU) ablative therapy for children with recurrent or relapsed solid tumors.
  Interventions: Device: Magnetic Resonance High Intensity Focused Ultrasound

INTERVENTIONS:
Device: Magnetic Resonance High Intensity Focused Ultrasound — MR-High intensity focused ultrasound (HIFU) is an ultrasound based technology which allows for non-invasive thermal ablation of tumors under the guidance of MR thermography.
  Other Names: MR-HIFU; HIFU; Philips Sonalleve

SUMMARY:
The purpose of this study is to determine if Magnetic Resonance guided High Intensity Focused Ultrasound ablative therapy is safe and feasible for children, adolescents, and young adults with refractory or relapsed solid tumors.

DETAILED DESCRIPTION:
Magnetic Resonance (MR)-guided high intensity focused ultrasound (HIFU) is an innovative technique that allows for non-invasive thermal ablation of tissue. Advantages over conventional local tumor control such as surgery, radiation, or radiofrequency are that MR-HIFU is completely non-invasive, non-ionizing, and enables ablation of large tumor volumes with avoidance of adjacent tissue injury. This study will evaluate the safety and feasibility of MR-HIFU ablative therapy in children, adolescents, and young adults with refractory or relapsed solid tumors that are located in bone or soft tissue in close proximity to bone. Patients ≤ 30 years of age with refractory or relapsed solid tumors with measurable target lesions that are located in bone or soft tissue in close proximity to bone are eligible. Tolerability will be defined during the 14 days following MR-HIFU ablation. Patients will continue to be followed for tumor response and secondary outcomes for up to one year post ablation treatment.

ELIGIBILITY:
Inclusion Criteria:

AGE: ≤ 30 years of age.

DIAGNOSIS:

Histologically confirmed malignant solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, germ cell tumors, and desmoid tumors.

TUMOR LOCATION: Target lesion(s) must be located in bone or soft tissue in close proximity to bone. Target lesions must be reachable within the normal safety margins of HIFU as specified in the instructions for use.

TARGET LESION(S): Radiographically evaluable or measurable solid tumor target lesion(s).

THERAPEUTIC OPTIONS:

Malignant Tumor: The patient's cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available. Curative therapy may include surgery, radiation therapy, chemotherapy, or any combination of these modalities.

PRIOR THERAPY:

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study.

No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.

Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry.

Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.

Biologic (anti-cancer agent): The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry.

Radiation therapy: The last dose of radiation to more than 25 % of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.

Stem Cell Transplantation. At least 2 months post-autologous stem cell transplant or at least 3 months post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease and on stable doses of immunosuppressive medications if required.

Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.

CONCURRENT THERAPIES:

No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) is permitted during HIFU treatment and post treatment follow up for tolerability (see section 3.3).

PERFORMANCE STATUS:

Patients > 16 years old must have a Karnofsky performance level ≥ 50%, and children ≤ 16 years old must have a Lansky performance level ≥ 50% (See Appendix I).

Patients who are unable to walk because of paralysis or motor weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.

* HEMATOLOGIC FUNCTION:

  1. Peripheral absolute neutrophil count (ANC) of ≥750/µL
  2. Platelet count ≥75,000/µL (may receive transfusions)
* RENAL FUNCTION: Age-adjusted normal serum creatinine OR a creatinine clearance ≥60 mL/min/1.73 m2.
* ADEQUATE PULMONARY FUNCTION: Defined as no dyspnea at rest, and a pulse oximetry >94% on room air if there is clinical indication for determination.
* Normal PT, PTT and INR < 1.5 x ULN (including patients on prophylactic anticoagulation)

Exclusion Criteria:

Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate the general anesthetic required for the procedure.

Implant or prosthesis or scar tissue within the path of the HIFU beam.

Target <1 cm from nerve plexus, spinal canal, bladder, bowel

Target in contact with hollow viscera

Lesion in the skull

Inability to undergo MRI and/or contraindication for MRI

Inability to tolerate stationary position during HIFU

Patients currently receiving other anticancer agents.

Patients currently receiving other investigational agents.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Toxicity | 28 days following ablative therapy
  Toxicity will be evaluated using CTCAEv4. Adverse events will be summarized descriptively with tabulations of adverse event type, severity, and relationship to study treatment.

SECONDARY OUTCOMES:
Disease response | Up to 1 year
  We will preliminarily define tumor response from MR-HIFU ablative therapy assessed according to a modified Response Evaluation Criteria in Solid Tumors (RECIST). We will also evaluate functional tumor response using FDG-PET post MR-HIFU ablative treatment for patients with PET avid target lesions.
Patient reported outcomes and quality of life measurements | Up to 1 year
  We will use a validated symptom distress scale and quality of life metrics pre- and post-therapy at scheduled intervals.
Immune Markers | Pre-treatment, 1 day post treatment, 7 days post treatment
  Changes in immune markers from baseline and post therapy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio